CLINICAL TRIAL: NCT01526278
Title: Pharmacokinetics of a Single Oral Dose of Maxmarvil® in Healthy Postmenopausal Women Without a Previous History of Fractures
Brief Title: Pharmacokinetics of Maxmarvil® in Healthy Postmenopausal Women
Acronym: YY_PK_2011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY_PK_2011
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Osteoporosis
Keywords: alendronate; Maxmarvil®
MeSH Terms: conditions — Osteoporosis | interventions — Maxmarvil; Alendronate; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maxmarvil® (Other): single-arm study
  Interventions: Drug: Maxmarvil®

INTERVENTIONS:
Drug: Maxmarvil® — Drug : Maxmarvil® 1tablet one time in clinical trial, PO medication
  Other Names: Alendronate 5mg + calcitriol 0.5 μg

SUMMARY:
This study will evaluate clinical safety and pharmacokinetics of Maxmarvil® in healthy postmenopausal women

DETAILED DESCRIPTION:
Pharmacokinetics of a single Oral Dose of Maxmarvil® in healthy postmenopausal women without a previous history of fractures

1. evaluation of Pharmacokinetics

   * Urine collection : Pre-dose(pre 1hour), post-dose 0~6 hour, 6~12 hour, 12~24 hour
   * Evaluation Variables : Aet
2. Evaluation of safety, pharmacodynamics

   * Adverse Event : check it every and frequently
   * Physical exam : screening, just before injection, post-dose 24 hour and post-study visit
   * Vital sign : screening, just before injection, post-dose 1 hour, 24 hour and post-study visit
   * Laboratory test : screening, post-dose 24hour

ELIGIBILITY:
Inclusion Criteria:

* Screening test in healthy postmenopausal women without a previous history of fracture
* Normal range in laboratory test arranged by principal investigator because of the character of medicine
* over 50kg, body weight is in ± 20% of ideal body weight Written concent by himself and following the protocol after understanding of the explained clinical trial

Exclusion Criteria:

* Subject who have taken something to induce and inhibit the drug metabolizing enzyme within 1 month like Barbiturate.
* Subject who have a history of drug abuse and got a positive in urine test for drug abuse.
* Subject who have taken a prescription only medicine or an oriental medicine within 2 weeks after first administration the clinical drug trial , taken a OTC within 1 week after first administration the clinical drug trial like some OTC including calcium, an antacids, multiple vitamin, mineral.
* Subject who have been chronic drinking(over 21 units/week) or can not stop drinking during the clinical trial.
* Subject who have smoked over 10 unit/day for 3months.
* Subject who have light or clear hypersensitivity reaction about OTC(aspirin, antibiotic medication) or bisphosphonates(alendronate)
* Subject who have got a disease about liver, kidney, neurology, respiratory, endocrine, hematooncology, cardiovascular, musculoskeletal, psychological or history of fracture within 12months or a tooth extraction within 6month
* Subject who have a history of gastrointestinal disease or stomach surgery without appendectomy, herniotomy having an effort the absorb of clinical drug trial.
* Subject who have a esophageal disease like esophagitis, esophageal ulcer, esophagus erosion, esophagorrhaphy, esophagostenosis, dysphagia.
* Subject who can not keep the sitting position for 30minutes
* Subject who is out of normal range of calcium concentration in blood (8.8 ~ 10.5 mg/dl)
* Subject who is hypotension(systolic blood pressure ≤ 90mmHg or diastolic blood pressure ≤ 50 mmHg ) or hypertension(systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100 mmHg ) in sitting position after rest 3 minutes
* join the other clinical trial within 2months after administration of the clinical drug trial.
* Subject who have donated whole blood within 2 months or plasma within 1 month.
* Subject who have a grapefruit and something including caffeine in close season(from 3 days before administration to discharge from the hospital )
* For the result of laboratory and the other reason subject is considered unsuitable by principal's decision

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
analysis of Alendronate concentrate | pre-dose, post dose 0-6hour, 6-12hour, 12-24hour
  If the CrCL value is less than 75%, it is considered that collected urine is not appropriate and collected urine is exclusived for analysis of pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: yoon-suk chung, MD,PhD, Principal Investigator — Ajou university hospotal
Locations (1):
- Ajou University Hospital, Suwon, South Korea